CLINICAL TRIAL: NCT05303857
Title: Randomized, Double-blind, Placebo Controlled, Parallel Group, Prospective Clinical Study to Analyse the Effect of Semaglutide on Vascular Structure and Function in Patients With Early Type 2 Diabetes
Brief Title: Analyse the Effect of Semaglutide on Vascular Structure and Function in Patients With Early Type 2 Diabetes
Acronym: SEMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Full Professor of Medicine, University Hospital Erlangen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRC2020SEMA
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: vascular structure; vascular function; GLP-1 analogue
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: randomized (1:1), double-blind, placebo controlled, parallel-group, prospective
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Baseline vascular function parameters will be obtained and the patient will be given semaglutide 1.34 mg/ml (SC, administered by personal injector, once weekly)
  Interventions: Drug: Semaglutide Pen Injector
- Placebo (Placebo Comparator): Baseline vascular function parameters will be obtained and the patient will be given placebo (SC, administered by personal injector, once weekly)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Pen Injector — Injection of the semaglutide once weekly
  Arms: Treatment
Drug: Placebo — Injection of placebo once weekly
  Arms: Placebo

SUMMARY:
This is a phase IV, randomized (1:1), prospective, double-blind, placebo controlled, parallel-group, single center study at the Clinical Research Unit (CRC) of the Department of Nephrology and Hypertension, with its two separate locations:

* Nürnberg, Kreuzburger Str. 2, 90471 Nürnberg, and
* Erlangen, Ulmenweg 18, 91054 Erlangen The main goal of the study is to demonstrate the effect of semaglutide on different vascular parameters of the macro- and microcirculation. The primary objective is to analyze the effect of semaglutide, compared to placebo on central (aortic) pulse pressure.

At least 90 patients will be randomized (1:1) and included (informed consent, intention to treat population) in order to obtain 80 fully evaluable subjects (per protocol population).

Patients will be simultaneously recruited from investigator's outpatient clinics, referring physicians, and advertisement in local newspapers, and social media. Those patients that appear to potentially fulfill the inclusion criteria will be invited to a screening visit (visit 1). After providing informed consent, patients will be tested for inclusion/exclusion criteria. Patients will provide a blood sample for laboratory testing. If the patient then fulfills inclusion criteria and in the absence of exclusion criteria, the patient will be enrolled into the trial, and the study visits will be scheduled. Randomization will take place at the latest one day prior to the study visit 2 (e.g. at the latest at visit 2a).

At visit 2 (2a and 2b), baseline vascular function parameters will be obtained and the patient will be given a SC injection of the study drug (either SC 0.25 mg semaglutide or SC placebo). After giving detailed instructions to the patient how to apply the injections, the patient will be advised to apply the injection once weekly. A safety visit will be conducted 1 week after first administration of study drug (visit 3). At visit 4 and 5, semaglutide will be up-titrated to 0.5 mg and 1.0 mg respectively. At visit 6, a safety visit will be conducted and the dose of semaglutide will be kept at 1.0 mg. After 16 weeks of treatment (visits 7a and 7b), testing of vascular function will be repeated. At visit 7b, a final close out visit will be performed to gather additional safety information.

DETAILED DESCRIPTION:
Diabetes mellitus type 2, considered at the beginning as a metabolic disorder, converts into a predominantly vascular disease, once its duration extends over several years or/and when additional cardiovascular risk factors like arterial hypertension coexist. Moreover, cardiovascular disease is the leading cause of death and complications in patients with type 2 diabetes. Recently, it has been demonstrated in a large longitudinal study that arterial stiffness is associated with higher risk of incident diabetes, independent of traditional risk factors. Increase in arterial stiffness appeared to even precede increase in fasting blood glucose. Moreover, we showed a reduced retinal capillary density in patients with prediabetes compared to patients with normal glucose metabolism (unpublished data). As a consequence, treatment of type 2 diabetes should focus not only on metabolic control but also on improving vascular structure and function, including endothelial function, the first stage of the atherosclerotic cascade.

In the last decade many studies have shown improved cardiovascular outcome in patients with type 2 diabetes treated with recently developed antidiabetic medication. The EMPA-REG Outcome trial evaluated the effect of a sodium-glucose cotransporter 2 inhibitor (empagliflozin) and have shown improved cardiovascular outcomes and lower rate of death from any cause in patients with type 2 diabetes who were at high risk for cardiovascular events. Similarly, in the LEADER trial first occurrence of death from cardiovascular causes, myocardial infarction, or stroke among patients with type 2 diabetes mellitus was lower with a glucagon-like peptide 1 analogue (liraglutide) than with placebo.

Semaglutide is another glucagon-like peptide 1 analogue with an extended half-life of approximately 1 week compared to liraglutide (efficacy and safety). Without any doubts, the large-scale prospective trial (SUSTAIN-6) demonstrating improved cardiovascular prognosis along with significant blood glucose reduction after treatment with semaglutide are very impressive and convincing, and this study fulfilled the regulatory guidance to establish cardiovascular safety of new therapies for type 2 diabetes. However this was primarily a non-inferior trial, although it demonstrated superiority with respect to the combined cardiovascular endpoint (p=0.02 for superiority). In the PIONEER-6 study conducted in patients with type 2 diabetes at least above 50 years with cardiovascular or chronic kidney disease or above 60 years and with cardiovascular risk factors, oral semaglutide proved cardiovascular safety. Other benefits of semaglutide in patient cohorts other than patients with type 2 diabetes has been described recently.

Several prospective studies reported a closer relation of organ damage with central (aortic) as opposed to peripheral (brachial) systolic blood pressure (BP), and central systolic BP was found to be independently associated with cardiovascular morbidity and mortality. In accordance, central pulse pressure has been repeatedly found to independently predict cardiovascular morbidity and mortality in various study cohorts. Further-more, prospective data have now been published showing that the forward and backward (reflected) wave amplitude predict independently cardiovascular complications. New advanced technology allows us to assess vascular parameters also under ambulatory conditions over 24 hours. Previously, we could demonstrate that the SGLT-2 inhibitors empagliflozin and dapagliflozin as well as the DPP-4 inhibitor saxagliptin improved parameters of vascular function and arterial stiffness and decreased central (aortic) pulse and systolic pressures (i.e. afterload of the left ventricle). Our results provided evidence for the concept that the better cardiovascular and renal outcomes observed with empagliflozin in the EMPA-REG Outcome Study are related to improved vascular function.

So far, there are no clinical data or an in-depth analysis of the effects on vascular function and stiffness after treatment with GLP-1 analogues, neither with liraglutide nor with semaglutide. In mice, semaglutide reduced the development of atherosclerosis by preventing the development of aortic plaques. Data supporting the concept that semaglutide improves vascular structure and function, including endothelial function are lacking, and our study aims at closing this knowledge gap by measuring various parameters of vascular remodeling and function at the same time thereby allowing us to delineate a complete profile of the vascular effects of semaglutide in the maco- and microcirculation. Such an approach is now in particular of relevance, since the European Medicines Agency (EMA) has already approved semaglutide s.c. (Ozempic) and semaglutide in an oral formula (Rybelsus) within the EU.

Our hypothesis is that in face of its impressive anti-diabetic effect semaglutide exerts beneficial effects on vascular structure and function, including endothelial function. Since the arterial pulse wave along the arterial tree is reflected at each bifurcation and thereby in particular at the ones of small arterioles, improvement in the vascular structure and function in microcirculation will also have profound consequences for the macrocirculation, as previously demonstrated, by lowering central pulse pressure and central systolic pressure both considered as valid and reliably measurable vascular parameters in the macrocirculation.

The main goal of the study is to demonstrate the effect of semaglutide on different vascular parameters of the macro- and microcirculation. The primary objective is to analyze the effect of semaglutide, compared to placebo on central (aortic) pulse pressure. Flow mediated vasodilation (FMD), an indicator of the integrity of endothelial function, is another parameter of the macrocirculation assessed in this study. Another parameter of the macrocirculation, assessed both in resting condition and 24-hours ambulatory conditions, in this study is pulse wave velocity (PWV), which is well known as an independent risk factor for cardiovascular morbidity and mortality. To analyze vascular remodeling processes in the microcirculation, we are measuring wall to lumen ratio of small retinal arterioles non-invasively in-vivo that reflects vascular remodeling of small arteries. Finally, only for a subgroup of up to 40 paitents parameters of the renal circulation including total renal perfusion, separate cortical and medullary renal perfusion and renal vascular resistance are measured using arterial spin labeling magnetic resonance imaging (ASL-MRI).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 75 years
* Diagnosis of type 2 diabetes mellitus: defined by fasting glucose ≥ 126 mg/dl or HbA1c ≥ 6,5 % or on oral single or dual blood glucose lowering medication (held constant for the last 3 months)
* HbA1c ≥ 7.0%
* Male and Female patients (females of child bearing potential must be using adequate contraceptive precautions)
* Females of childbearing potential or within two years of the menopause must have a negative urine pregnancy test at screening visit
* Informed consent (§ 40 Abs. 1 Satz 3 Punkt 3 AMG) has to be given in written form

Exclusion Criteria:

* Any other form of diabetes mellitus than type 2 diabetes mellitus
* Use of insulin, sulfonylurea or GLP-1 analogue within the past 3 months
* Patients with more than two oral blood glucose lowering medication
* HbA1c ≥ 10.5%
* Body mass index > 40 kg/m²
* Fasting plasma glucose > 240 mg/dl
* Any form of diabetic retinopathy, macular oedema
* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m²
* Acute or chronic pancreatitis
* Uncontrolled arterial hypertension (BP ≥ 180/110 mmHg)
* Any history of stroke, transient ischemic attack, instable angina pectoris, or myocardial infarction within the last 3 months prior to study inclusion
* Congestive heart failure (CHF) NYHA stage III and IV
* Drug or alcohol abuses
* Pregnant or breast-feeding patients

Subset of patients receiving ASL-MRI, exclusion criteria-

Patients with contraindications to MRI, including:

* Brain aneurysm clip
* Implanted neural stimulator
* Implanted cardiac pacemaker or defibrillator, or presence of intracardiac wires
* Prosthetic heart valves
* Cochlear implant
* Ocular foreign bodies that might be ferromagnetic (e.g., metal shavings)
* Other implanted medical devices (e.g., insulin pumps)
* Metal shrapnel or bullets still in the body
* Severe claustrophobia
* Tattoos (as determined by the Investigator and Imager)
* Weight in excess of MRI machine capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Central (aortic) pulse pressure assessed by Sphygmocor XCEL | 16 weeks
  The primary objective of the study is to analyze the effect of semaglutide, compared to placebo, on:
  central (aortic) pulse pressure after 16 weeks of treatment from baseline

SECONDARY OUTCOMES:
Central (aortic) systolic pressure assessed by Sphygmocor XCEL | 16 weeks
  change of central (aortic) systolic pressure after 16 weeks of treatment from baseline
Augmentation pressure assessed by Sphygmocor XCEL | 16 weeks
  change of augmentation pressure after 16 weeks of treatment from baseline
Augmentation index (cAIX@75) assessed by Sphygmocor XCEL | 16 weeks
  change of augmentation index (cAIX@75) after 16 weeks of treatment from baseline
Forward wave amplitude assessed by Sphygmocor XCEL | 16 weeks
  change of forward wave amplitude after 16 weeks of treatment from baseline
Backward wave amplitude assessed by Sphygmocor XCEL | 16 weeks
  change of backward wave amplitude after 16 weeks of treatment from baseline
Outer diameter of small retinal arterioles assessed by Scanning laser Doppler flowmetry | 16 weeks
  change of outer diameter of small retinal arterioles after 16 weeks of treatment from baseline
Inner diameter of small retinal arterioles assessed by Scanning laser Doppler flowmetry | 16 weeks
  change of inner diameter of small retinal arterioles after 16 weeks of treatment from baseline
Wall to lumen ratio of small retinal arterioles assessed by Scanning laser Doppler flowmetry | 16 weeks
  change of wall to lumen ratio of small retinal arterioles after 16 weeks of treatment from baseline
Flow-mediated Vasodilation (FMD) of the brachial artery assessed by UNEX EF | 16 weeks
  change of FMD of the brachial artery after 16 weeks of treatment from baseline
Pulse wave velocity assessed by Sphygmocor XCEL | 16 weeks
  change of pulse wave velocity after 16 weeks of treatment from baseline
24-h ambulatory BP (brachial and central) assessed by Mobil-O-Graph® | 16 weeks
  change of 24-h ambulatory BP (brachial and central) after 16 weeks of treatment from baseline
24-h ambulatory vascular parameter assessed by Mobil-O-Graph® | 16 weeks
  change of 24-h ambulatory vascular parameter (pulse wave velocity) from baseline
24-h ambulatory vascular parameter assessed by Mobil-O-Graph® | 16 weeks
  change of 24-h ambulatory vascular parameter (central pulse pressure, central systolic pressure) from baseline
Renal perfusion of both kidneys assessed by Arterial Spin Labeling MRI | 16 weeks
  change of renal perfusion (total, cortical, medullary) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Roalnd E Schmieder, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No